CLINICAL TRIAL: NCT03381924
Title: Effectiveness of a Group Educational Intervention in Patients With Migraine: a Randomised Controlled Trial
Brief Title: Educational Intervention in Patients With Migraine
Acronym: M01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Iñaki Aguirrezabal Bazterrica, General Practitioner, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIGRAINE01
Record Dates: First submitted 2017-12-14; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Migraine
Keywords: Migraine disorders; Educational models; Neuroscience
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Neuroscience-based information on the neurophysiology of pain and migraine were provided with audio-visual support.
  Interventions: Other: Educational programme
- Control group (Placebo Comparator): Routine clinical practice
  Interventions: Other: Routine clinical practice

INTERVENTIONS:
Other: Educational programme — In each session, neuroscience-based information on the neurophysiology of pain and migraine were provided with audio-visual support.
  Arms: Intervention group
Other: Routine clinical practice — Patients allocated to the control group will only receive the drugs used in the habitual clinical practice
  Arms: Control group

SUMMARY:
Introduction: Despite the numerous pharmacological treatment options available for migraine attacks and for the prevention of thereof, less than 30% of patients with migraine are highly satisfied with their current treatment.

In recent decades, there has been a radical change in the way we view pain, thanks to developments in neuroscience. It is currently considered that pain does not originate in the peripheral nociceptors, but rather in a network of brain regions (the pain neuromatrix), the synchronous activation of which is necessary and sufficient to generate the perception of pain. Migraine may be the expression of this exaggerated perception of threat, a perception that, from a cultural learning perspective, it may be possible to modify by adjusting beliefs and behaviours that favour the onset of an attack.

The aim of this study was to assess the effectiveness of a group educational intervention about concepts of pain neuroscience, in the management of migraine, compared to routine medical interventions, in primary care health centres of Alava.

DETAILED DESCRIPTION:
The aim of this study was to assess the effectiveness of a group educational intervention about concepts of pain neuroscience, in the management of migraine, compared to routine medical interventions, in primary care health centres of Alava.

After recruitment, patients were interviewed by the research team members in charge of the assessments. In these interviews, data were collected on the following: demographic characteristics, beliefs regarding migraine, coping strategies for migraine attacks, the MIDAS questionnaire (16), medication taken, work leave, emergency department attendances and limitation of daily activities due to migraine, during the previous 3 months.

Subsequently, we carried out further assessments over the telephone after 3, 6 and 12 months. Very few studies assessing preventive treatments for migraine have performed assessments 12 months after initiating prophylactic treatment, most having followed-up patients for 6 months at most. We believe, however, it is necessary to continue assessments for at least 1 year to properly test the efficacy of treatment for chronic illnesses like migraine. The individuals carrying out the assessment were blinded to group allocation. The clinical follow-up was the same for both groups, the only difference in their management being the educational intervention itself.

ELIGIBILITY:
Inclusion Criteria:

* Belong to one of these health centres of primary care: San Martín, Sansomendi, Lakuarriaga, Gazalbide and Zabalgana,
* Diagnosed with migraine (ICD-9-CM Diagnosis Code 346) who had at least one migraine attack every month despite treatment.

Exclusion Criteria:

* We excluded patients with mental illness, cognitive impairment or language deficits that might hinder completion of follow-up and patients that would not be able to attend to all the sessions of the intervention or had received training as part of the previous pilot study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Migraine-related disability given by the MIDAS score | 12 months
  The sum of responses to five questions on days missed or with reduced productivity at work/school, at home and in leisure activities.I If patients has reduced the score in MIDAS scale by at least the 50% of the baseline score, we consider that the patient has responded to the treatment.

SECONDARY OUTCOMES:
Intensity and frequency of the pain | 12 months
  Measured using the two supplementary questions of the MIDAS, the two supplementary questions of the MIDAS. If patients has reduced the score in MIDAS scale by at least the 50% of the baseline score, we consider that the patient has responded to the treatment.
Degree to which activities of daily life were limited by migraine | 12 months
  Measured using an ad hoc scale with six possible answers: not at all, very little, little, quite a lot, a lot, and totally.
costs associated with migraine-related treatment | 12 months
  Both preventive medication and medication for treating migraine attacks

CONTACTS AND LOCATIONS:
Overall Officials: IÑAKI AGUIRREZABAL, Principal Investigator — Basque Health Service
Locations (1):
- Iñaki Aguirrezabal Bazterrica, Vitoria-Gasteiz, Alava, Spain